CLINICAL TRIAL: NCT00203905
Title: A Randomized Phase II Study of Concomitant Chemoradiotherapy With 5-Fluorouracil/Hydroxyurea Compared to FHX Plus Bevacizumab for Intermediate Stage and Selected Stage IV Cancers of the Head and Neck
Brief Title: A Study of Chemoradiotherapy for Intermediate Stage/Selected Stage IV Cancers of the Head and Neck
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 12652A
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2014-01

CONDITIONS: Head and Neck Cancer
Keywords: Head and Neck Cancer
MeSH Terms: conditions — Head and Neck Neoplasms | interventions — Fluorouracil; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Hydroxyurea at 500 mg PO q 12 hours x 6 days (11 total doses); Infusion of 5-FU (600 mg/m2/day x 5 days [120 hours]
  Interventions: Drug: 5-Fluorouracil, Hydroxyurea-[FHX]
- B (Experimental): Bevacizumab: 10 mg/kg will be given as a 90-minute infusion
  Interventions: Drug: 5-Fluorouracil, Hydroxyurea-[FHX], Bevacizumab

INTERVENTIONS:
Drug: 5-Fluorouracil, Hydroxyurea-[FHX], Bevacizumab — Hydroxyurea at 500 mg PO q 12 hours x 6 days; Bevacizumab at 10 mg/kg as a 90-minute infusion; Infusion of 5-FU (600 mg/m2/day) X 5 days (120 hours)
  Arms: B
Drug: 5-Fluorouracil, Hydroxyurea-[FHX] — Hydroxyurea at 500 mg PO q 12 hours x 6 days; Infusion of 5-FU (600 mg/m2/day) X 5 days (120 hours)
  Arms: A

SUMMARY:
The primary objective of the study is to evaluate time to progression in eligible patients with cancer of the oral cavity, pharynx, larynx, paranasal sinuses, and cervical esophagus when treated with the concomitant chemoradiotherapy regimen of bevacizumab/5-fluorouracil (5-FU)/hydroxyurea/radiation therapy (B-FHX) in comparison to 5-fluorouracil hydroxyurea (FHX) alone.

DETAILED DESCRIPTION:
In this study, we intend to explore the feasibility and the effects of adding bevacizumab to Fl-TX in patients with intermediate stage head and neck cancer and selected patients with stage IV disease. As mentioned previously, although single modality therapy (surgery or radiotherapy alone) is often used to treat patients with Stage II head and neck malignancies, with substantial success, still there is a sizeable group of patients (approximately 30% or 40%) who fail these treatments, and represent with locoregional recurrences which are much more difficult to treat. Furthermore, the common use of radical surgery in many instances leads to loss of organ function.

Based on this knowledge, we feel that it is justifiable to include stage II patients (T2NO) in combined chemoradiation studies. Our extensive experience using chemoradiotherapy in patients with regionally advanced non-metastatic Stage 4 cancers of the head and neck area suggests that selected patients with low nodal status (Nondisease) including those with T4 primaries (i.e. T4 NO MO and T4 Nl MO) have a lower risk of distant failure than patients that present with higher nodal status (N2 and N3 disease). Aggressive combined locoregional therapies such as the one that will be administered in the study, are in our opinion appropriate for this group of patients as they address the major concern which is locoregional failure.

The primary goal of the study is exploration of the pharmacodynamic effects of bevacizumab (10 mg/kg) on appropriate markers of angiogenesis in tumor tissue in comparison to a non-bevacizumab containing chemoradiation regimen (FHX alone). These results will be correlated with a number of clinical endpoints including rapidity of clinical response, locoregional control rates, time to progression, need of salvage surgery, overall survival and measures of QOL and organ function. The predictive and prognostic value of specific molecular markers in patients with HNC will also be evaluated. In order to shorten the total duration of treatment without affecting the total administered dose, we have modified our traditional radiation schedule in FHX to include two treatment daily fractions as opposed to one. This modification will allow for the completion of all treatment in 4 to 5 cycles as opposed to the traditional 6 to 7 cycles. Given this modification in the radiation schedule, we considered it prudent to include a control arm (modified FHX) in addition to B-FHX, within a randomized design. The control arm will also help with the interpretation of the results obtained with the measurement of the correlative markers of angiogenesis.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have stage II-III (carcinoma of head and neck, including oral cavity, pharynx, larynx, paranasal sinuses and cervical esophagus). Selected patients with stage disease (T will also be considered for enrolment). Therapy is given with curative intent. Patients with clinical N2 or N3 disease are excluded.
* Prior to entry in the study the resectability and standard treatment options for each patient will be determined during a joint evaluation by a team composed of an attending surgeon, a radiation oncologist and a medical oncologist. In addition the timing and feasibility of initial organ preserving surgery will be determined in each patient prior to therapy at the discretion of the treating surgeon. Salvage surgery and neck dissection will be allowed for suspicious or evident residual disease at the completion of the treatment regimen.
* Measurable disease is not required.
* Patients must have a histologically or cytologically confirmed diagnosis of carcinoma of the head and neck.
* No prior exposure to chemotherapy or radiotherapy for a malignancy of the head and neck.
* Patients must have ECOG performance status of 0-2.
* Age 18 years of age and older.
* Patients must have normal organ and bone marrow function.

Exclusion Criteria:

* Receiving any other investigational agents
* Recent (within 6 months) myocardial infarction, New York Heart Association (NYHA) - Class H or greater congestive heart failure, serious cardiac arrhythmia requiring medication, or Grade II or greater peripheral vascular disease within 1 year prior to treatment in the study
* Serious, non-healing wound, ulcer, or bone fracture.
* History of recurrent or chronic deep vein thrombosis or pulmonary embolus
* History of CNS disease (including CNS involvement from primary cancer) or hemorrhagic or thrombotic stroke within the last 6 months
* Uncontrolled hypertension
* Evidence of bleeding diathesis or coagulopathy
* History of hemoptysis
* Anatomic lesion that increases the risk of serious hemorrhage (e.g. invasion of a major vessel by tumor).
* History of other disease, metabolic dysfunction, physical examination finding, or clinical laboratory finding giving reasonable suspicion of a disease or condition that contraindicates the use of an investigational drug or that might affect the interpretation of the results of the study or render the subject at high risk from treatment complications.
* Current ongoing treatment with any dose of warfarin or its equivalent.
* Major surgical procedure or significant traumatic injury within 28 days prior to Day 0.
* Fine needle aspirations, indwelling catheter placement, or significant traumatic injury within 7 days prior to Day 0
* Anticipation of need for major surgical procedure during the course of the study.
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to rhuMAb VEUF or other agents used in the study.
* History of a concurrent malignancy or a history of a prior malignancy within the past 3 years.
* Pregnant women
* HIV-positive patients receiving combination anti-retroviral therapy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2004-01; Primary Completion 2007-11 (Actual); Study Completion 2008-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the time to progression free survival in patients with cancer of the oral cavity, pharynx, larynx, paranasal sinuses, and cervical esophagus when treated with the concomitant chemoradiotherapy regimen | From randomization until disease progression or death from any cause

SECONDARY OUTCOMES:
To explore the pharmacodynamic changes induced on selected markers of angiogenesis by the addition of bevacizumab to FHX and compare them to those induced by FHX alone | Baseline, week 2, and completion of therapy

CONTACTS AND LOCATIONS:
Overall Officials: Everett Vokes, M.D., Principal Investigator — University of Chicago
Locations (1):
- The University of Chicago, Chicago, Illinois, United States